CLINICAL TRIAL: NCT00002538
Title: LAPAROSCOPIC STAGING IN PATIENTS WITH INCOMPLETELY STAGED CANCERS OF THE OVARY
Brief Title: Laparoscopic Staging in Patients With Ovarian, Fallopian Tube, or Other Primary Abdominal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: GOG-9302; CDR0000078530
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: laparoscopic surgery

SUMMARY:
RATIONALE: Laparoscopic staging may help doctors plan more effective treatment for ovarian, primary fallopian tube, and primary abdominal cancers.

PURPOSE: Phase II trial to study the effectiveness of laparoscopic staging in patients with ovarian, primary fallopian tube, or primary abdominal cancers who have not undergone complete staging.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of laparoscopic staging of patients with incompletely staged ovarian, primary fallopian tube, and primary peritoneal cancers. II. Assess the adverse effects associated with this technique.

OUTLINE: Surgery. Laparoscopy with cytologic examination and lymph node sampling followed, if feasible, by surgical resection.

PROJECTED ACCRUAL: Up to 50 patients will be accrued over approximately 2 years. If more than 4 evaluable patients cannot complete surgery, the study will be closed.

ELIGIBILITY:
DISEASE CHARACTERISTICS: One of the following incompletely staged malignancies: Ovarian cancer of any cell type Primary fallopian tube carcinoma Primary peritoneal carcinoma No clinical evidence of metastases to abdominal organs, the adnexa, or retroperitoneal lymph nodes on CT with contrast or at prior abdominal surgery No metastases on chest x-ray No contraindications to laparoscopy, i.e.: No bowel obstruction No ileus No peritonitis No excessive obesity as indicated by a Quetelet Index over 35 (weight in kg/height in sqm) No diaphragmatic hernia on chest x-ray No grade 2 heart toxicity

PATIENT CHARACTERISTICS: Age: Adult Performance status: GOG 0 or 1 Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no more than 1.5 mg/dL AST no more than 3 times normal Renal: Creatinine no more than 2.0 mg/dL Other: No second malignancy except nonmelanomatous skin cancer Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior or concomitant chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior or concomitant abdominal or pelvic radiotherapy Surgery: No prior retroperitoneal surgery No more than 10 weeks since initial abdominal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1993-09; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick M. Spirtos, MD, Study Chair — Women's Cancer Center - Palo Alto
Locations (11):
- United States (11):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Women's Cancer Center, Palo Alto, California
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania

REFERENCES:
- [Background] Spirtos NM, Eisekop SM, Boike G, Schlaerth JB, Cappellari JO. Laparoscopic staging in patients with incompletely staged cancers of the uterus, ovary, fallopian tube, and primary peritoneum: a Gynecologic Oncology Group (GOG) study. Am J Obstet Gynecol. 2005 Nov;193(5):1645-9. doi: 10.1016/j.ajog.2005.05.004. PMID 16260204